CLINICAL TRIAL: NCT06241443
Title: The Impact of Simulation-Based Education on Positive Birth Perception and Natural Birth Approach
Brief Title: Nursing Students & Positive Birth Perception & Simulation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ege University (Other)
Responsible Party: Principal Investigator, sümeyye bakır, doctoral student/research assistant, Ege University
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Health Services Research
Other Study IDs: E.1161
Record Dates: First submitted 2024-01-27; First posted 2024-02-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2024-01

CONDITIONS: Childbirth Problems
Keywords: childbirth experience; nursing students; simulation-based education; positive birth

STUDY DESIGN:
Intervention Model Description: prospective, parallel, randomized, controlled quasi-experiment
Who Masked: Participant
Masking Description: The students who participated in the research were unaware of their assigned group.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- hybrid simulation (Experimental): These students participated in a natural birth approach scenario with a hybrid simulation (n=28).
  Interventions: Other: hybrid simulation
- video-modeling group (Active Comparator): The students in this group participated in a video modeling education (n=28).
  Interventions: Other: video-modeling

INTERVENTIONS:
Other: hybrid simulation — During the hybrid simulation, a student and a standardized patient participated. The patient wore a wearable pregnancy model. Before the start of the "Natural Birth Approach Scenario, a pre-briefing session was conducted. The student's performance during the simulation was recorded on video, and each simulation lasted approximately 30 minutes. After the simulation, a debriefing session was held with the student, and feedback was given. Scales were used to evaluate the implementation of the practices.
  Arms: hybrid simulation
Other: video-modeling — The students in the group had the opportunity to learn through an educational video that followed the "Natural Birth Approach Scenario." Afterward, they put their knowledge into practice and were evaluated using the Birth Approach Clinical Skills Guide. A feedback session followed the practice session. Finally, they were assessed using scales to measure their performance.
  Arms: video-modeling group

SUMMARY:
The study aimed to investigate the impact of simulation-based training on nursing students' perception of positive birth and natural birthing approaches.

DETAILED DESCRIPTION:
This study aimed to determine whether simulation-based training could improve the perception of positive birth and natural birthing approaches among fourth-year nursing students. The study used a randomized controlled quasi-experimental design with pre-test and post-test. The intervention group received hybrid simulation, while the other received video-modeling training. The study used several tools to assess the impact of the training, including the Demographic Information Form, Natural Birth Approach Questionnaire, Student Satisfaction and Confidence in Learning Scale, Satisfaction with Education Methods Questionnaire, and Natural Birth Approach Clinical Skills Guide.

ELIGIBILITY:
Inclusion Criteria:

* The voluntarily agree to participate in the study Not having experience with simulation Being a 4th year nursing undergraduate student not working as a nurse

Exclusion Criteria:

* During the study, participants must complete all forms, attend all theoretical training, and remain in the study until completion.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2022-09-20 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-06-20 (Actual)

PRIMARY OUTCOMES:
Natural Birth Approach Questionnaire | change from before implemention and 4th week of after practice
  The researchers developed a measurement tool to assess students' knowledge, opinions, and approaches to natural birth. The tool uses a scoring system where correct statements receive one point and incorrect statements receive zero points. The total score ranges from 0 to 100 points.
students' self-confidence and satisfaction | through simulation practices completion, an average of 5 weeks
  It is a scale published by the National League for Nurses (NLN) to measure students' attitudes and beliefs about simulation.The highest score that can be obtained from the scale is 65 and the lowest score is 13.
education methods satisfaction | through simulation practices completion, an average of 5 weeks
  It evaluates the degree of contentment of the student with the teaching methodology implemented.In evaluating the satisfaction with training methods, students are scored from 20 to 80.
Natural Birth Approach Skills | through simulation practices completion, an average of 5 weeks
  The researchers developed a checklist to assess skills. Each item was evaluated on a 3-point scale indicating inadequacy, partial sufficiency, or sufficiency. The checklist consists of 21 items. The total score ranges from 21 to 63 points.

CONTACTS AND LOCATIONS:
Overall Officials: sümeyye bakır, master, Principal Investigator — Ege University
Locations (1):
- Ege Univesity, Izmir, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes
The researchers intend to publish the study as an article
Supporting Information: Study Protocol
Time Frame: from January 2025
Access Criteria: the article is planned to be published as open access

REFERENCES:
- [Background] Dunbar-Reid K, Sinclair PM, Hudson D. Advancing renal education: hybrid simulation, using simulated patients to enhance realism in haemodialysis education. J Ren Care. 2015 Jun;41(2):134-9. doi: 10.1111/jorc.12112. Epub 2015 Jan 29. PMID 25631292
- [Result] Bakke E, Oseth EH, Fofanah T, Sesay I, van Duinen A, Bolkan HA, Westendorp J, Lonnee-Hoffmann R. Vacuum births and barriers to its use: An observational study in governmental hospitals in Sierra Leone. BMJ Open. 2022 Nov 22;12(11):e060773. doi: 10.1136/bmjopen-2022-060773. PMID 36414288
- [Result] Duff J, Kardong-Edgren S, Chang TP, Elkin RL, Ramachandra G, Stapleton S, Palaganas JC, Kou M, Gross IT. Closing the gap: a call for a common blueprint for remote distance telesimulation. BMJ Simul Technol Enhanc Learn. 2021 Apr 12;7(4):185-187. doi: 10.1136/bmjstel-2021-000875. eCollection 2021. PMID 35516822